CLINICAL TRIAL: NCT00235521
Title: Comparison of Inhaled Nitric Oxide With Aerosolized Iloprost (Ventavis®) for Treatment of Pulmonary Hypertension in Children After Cardiopulmonary Bypass Surgery
Brief Title: Iloprost-Study: Comparison of Nitric Oxide to Iloprost (Ventavis) for Treatment of Pulmonary Hypertension in Children After Cardiopulmonary Bypass Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Heidelberg University (Other)
Responsible Party: Principal Investigator, Matthias Gorenflo, Prof. Dr. med., Heidelberg University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Iloprost-Study
Record Dates: First submitted 2005-10-06; First posted 2005-10-10 (Estimated); Last update posted 2012-12-12 (Estimated); Status verified 2012-12

CONDITIONS: Pulmonary Hypertension
Keywords: Pulmonary hypertension; Cardiac Surgery; Children; Pediatric Patients; Iloprost; NO; nitric oxide; Pulmonary hypertension after cardiac surgery in pediatric patients, 0 - 2 years old
MeSH Terms: conditions — Hypertension, Pulmonary

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: aerosolized iloprost

SUMMARY:
Inhaled nitrous oxide (iNO) will be compared to aerosolized iloprost (ILO) in pediatric patients after cardiac surgery with pulmonary hypertension. The hypothesis is that iloprost is more effective in preventing pulmonary hypertensive crises.

DETAILED DESCRIPTION:
Investigators, Study Sites: Single-center trial at the Department of Pediatric Cardiology, Department of Cardiac Surgery and Department of Anesthesiology, University Medical Center, Heidelberg, Germany Exploratory proof of concept study (Investigator initiated trial)

Indication: Postoperative pulmonary hypertension in infants and children undergoing cardiopulmonary bypass surgery for intracardiac repair of left-to-right shunt

Objectives: To compare the efficacy of aerosolized iloprost with inhaled nitric oxide to prevent postoperative pulmonary hypertensive crises

Design: Exploratory, open label, randomized study with parallel-group design;

Duration of observation: 72 hours

Population: Infants older than 4 weeks and children less than 18 months of age presenting with left-to-right shunt and increased pulmonary blood flow. Inclusion will be independent on the presence or absence of preoperative pulmonary hypertension

Sample Size:

* 20 patients: inhaled nitric oxide (iNO) - group;
* 20 patients: aerosolized iloprost (ILO) -group

Treatment:

* Both groups: controlled ventilation, sedation, analgetics, inotropic substances as required, standardized intensive care treatment.
* iNO - group: concentration of iNO at 10 ppm; administered by mechanical ventilation.
* ILO - group: aerosolized Iloprost at a dose of 0,5 µg/kg body weight (12x / 24h), administered by ultrasound nebulizer.

Efficacy Parameters: Occurrence of "minor" or "major" pulmonary hypertensive crises (PHTC)

Safety Parameters: Arterial blood pressure, oxygen saturation, complete blood count

Statistical Procedures: All analyses in this exploratory trial are descriptive, giving confidence intervals for differences between treatment groups.

Primary analysis variable: Rate of occurrence of "major" or "minor" pulmonary hypertensive crises

Secondary variables: Presence of hours of pulmonary hypertension, Duration of mechanical ventilation

ELIGIBILITY:
Inclusion Criteria:

* Informed consent by parents or legal representatives
* Age: Infants older than 4 weeks of age and children less than 1½ years of age.
* Presence of a left-to-right shunt with increased pulmonary blood flow. The specific defects that will be present are:

  * Aortopulmonary (AP) - Window
  * Atrioventricular septal defect (AVSD)
  * Double outlet right ventricle (DORV)
  * Total anomalous pulmonary venous drainage (TAPVD)
  * Truncus arteriosus
  * Ventricular septal defect (VSD)
* Presence of postoperative PH immediately after intracardiac repair:

  * Patients will be enrolled if mean PAP after intracardiac repair exceeds 25 mmHg after weaning from CPB.

Exclusion Criteria:

* Specific cardiac defects:

  * Atrial septal defect (ASD)
  * Cyanotic congenital heart disease
  * Univentricular atrio-ventricular - connexion
  * Valvular or subvalvular pulmonary or aortic stenosis
* Specific circumstances:

  * Emergency cardiac surgery
  * Children presenting with infection after cardiac surgery
  * Infants on extracorporeal membrane oxygenation (ECMO) before cardiac surgery
  * Infants/children treated with epoprostenol
* Concomitant diseases:

  * Systemic arterial hypertension
  * Renal failure
  * Diabetes mellitus
  * Known bleeding disorders (known disorders of blood coagulation and hemostasis)
  * Infection during the first 24 hours after cardiac surgery

Max Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 15 (Actual)
Dates: Start 2005-05; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Number of pulmonary hypertensive crises (major and/or minor)

SECONDARY OUTCOMES:
Treatment with aerosolized ILO is equally effective as iNO in reducing the pulmonary artery pressure (PAP) within the first 72 hours after cardiopulmonary bypass surgery (CPB)
Patients treated with aerosolized ILO can be weaned earlier from mechanical ventilation than patients on iNO treatment
Patients treated with aerosolized ILO show the same in-hospital mortality as patients treated with iNO

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Gorenflo, MD, PhD, Principal Investigator — Heidelberg University
Locations (1):
- University of Heidelberg, Medical Faculty, Department of Pediatric Cardiology, Heidelberg, Germany